CLINICAL TRIAL: NCT01717066
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Study to Evaluate the Efficacy and Safety of Ginsenoside Rg3 Capsule in Prevention of Postoperative Recurrence of Hepatocellular Carcinoma
Brief Title: the Efficacy and Safety of Ginsenoside Rg3 Capsule in Prevention of Postoperative Recurrence of Hepatocellular Carcinoma
Acronym: Rg3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ShenFeng (Other)
Collaborators: Huazhong University of Science and Technology (Other); Shanghai Zhongshan Hospital (Other); Sun Yat-sen University (Other); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor-Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EHBH-RCT-2011-002
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Stage I Hepatocellular Carcinoma; Stage II Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; ginsenoside Rg3
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the ginsenoside Rg3 (Experimental): 320 HCCs,the ginsenoside Rg3 capsule,4-8 weeks after surgery, will be taken, 2 capsules, BID, 8 weeks as one cycle, continue taking it until the tumor recurs or until the end date of the study for patients without recurrence
  Interventions: Drug: the ginsenoside Rg3
- the placebo (Placebo Comparator): 160 HCCs as control group with patients who don't receive any adjuvant therapy after liver resection, to compare with the treatment group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: the ginsenoside Rg3
  Other Names: Shen Yi capsule
  Arms: the ginsenoside Rg3
Drug: Placebo
  Arms: the placebo

SUMMARY:
Using the subject with hepatocellular carcinoma in the conventional therapy to evaluate the efficacy and safety of ginsenoside Rg3 (20mg BID) and placebo in prevention and treatment of postoperative recurrence of liver cancer,respectively

DETAILED DESCRIPTION:
1. Randomized, double-blind, multi-center, placebo-controlled, parallel-group;
2. Subject population: patients undergone radical resection of hepatocellular carcinoma;
3. Active drug group:

Ginsenoside Rg3 group: general treatment + ginsenoside Rg3 Control group (placebo group): general treatment + placebo 4.Method of group assignment: 5research centers, central-block-stratified randomization, a ratio of active drug group to control group: 2:1 5.Dose and mode of administration: Ginsenoside Rg3 group: ginsenoside Rg3 20mg BID, two months as one cycle, continue until recurrence occurs Placebo Group: placebo, 2 capsules, BID, continue until recurrence occurs 6.Study period: Screening phase: screening for enrollment within 8 weeks after the radical resection Follow up: review every 2-3 months following the surgery Post-trial investigation: within 28 days after the trial is ended or the recurrence occurs

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old,male and female
* Mainly based on the criteria for liver cancer TNM stage I and II (edition 7) and BCLC stage A, the following needs to be satisfied:

  1. individual tumor larger than or equal to 2 cm and smaller than or equal to 10 cm in the maximum diameter
  2. multiple tumors with no more than three tumors
  3. No macroscopic tumor embolus
* ECOG performance state is 0-1
* Child-Pugh grade is A
* The clinical review confirms the absence of recurrence within 8 weeks before the enrollment
* Sign the informed consent

Exclusion Criteria:

* Pregnant and breast-feeding women
* Patients with severe diseases in the brain, heart,lungs, kidneys and hematological system
* Patients who have received other anti-tumor therapies before the surgery (including liver transplantation, TACE, local tumor ablation, chemotherapy, radiotherapy, molecular targeted therapy and other anti-tumor therapy)
* DDS chemotherapy pump placed in the portal vein during the surgery
* Patients who are participating in other drug trials
* Patients known or suspected to be allergic to ginsenoside, with a history of allergy to biological preparations, allergic constitution or currently in an allergic state;
* With active severe clinical infection
* Epilepsy episode which needs drug therapy
* With a history of allotransplantation;
* With a previous history of tumor in other systems, but except for:

  1. Carcinoma in situ of cervix
  2. Basal cell carcinoma after treatment,Superficial bladder cancer (Ta, Tis and T1
  3. Any cancer after curative treatment no less than three years ago
* Patients with signs or a history of bleeding diathesis
* Patients currently receiving kidney dialysis
* A history of bleeding in the gastrointestinal tract within 30 days, or severe gastroesophageal varices with red signs; with a history of gastroesophageal variceal hemorrhage
* Recurrent HCC
* Patients unable to take drug orally
* Patients inappropriate to participate in the trial upon the investigator's judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
time to recurrence | 1,2,3 years
  the interval between the initial hepatectomy and date of diagnosis of recurrent HCC

SECONDARY OUTCOMES:
overall survival | 1,2,3 years
  the interval between the date of the initial hepatectomy and the date of death or last follow-up

OTHER OUTCOMES:
side effect | eighteen months
  the adverse reactions of the application of ginsenoside Rg3,for example:severe dry pharynx

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, MD,PhD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital
Locations (5):
- China (5):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Tumor Hospital,Sun Yat-san University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Tongji Hospital,Huazhong University of Science ＆ Technology, Wuhan, Hubei
  - Zhongshan hospital,Fudan University, Shanghai

REFERENCES:
- [Background] Yue PY, Wong DY, Wu PK, Leung PY, Mak NK, Yeung HW, Liu L, Cai Z, Jiang ZH, Fan TP, Wong RN. The angiosuppressive effects of 20(R)- ginsenoside Rg3. Biochem Pharmacol. 2006 Aug 14;72(4):437-45. doi: 10.1016/j.bcp.2006.04.034. Epub 2006 May 12. PMID 16793023
- [Background] Liu TG, Huang Y, Cui DD, Huang XB, Mao SH, Ji LL, Song HB, Yi C. Inhibitory effect of ginsenoside Rg3 combined with gemcitabine on angiogenesis and growth of lung cancer in mice. BMC Cancer. 2009 Jul 23;9:250. doi: 10.1186/1471-2407-9-250. PMID 19624862
- [Background] Zhang Q, Kang X, Yang B, Wang J, Yang F. Antiangiogenic effect of capecitabine combined with ginsenoside Rg3 on breast cancer in mice. Cancer Biother Radiopharm. 2008 Oct;23(5):647-53. doi: 10.1089/cbr.2008.0532. PMID 18999937
- [Background] Xu TM, Cui MH, Xin Y, Gu LP, Jiang X, Su MM, Wang DD, Wang WJ. Inhibitory effect of ginsenoside Rg3 on ovarian cancer metastasis. Chin Med J (Engl). 2008 Aug 5;121(15):1394-7. PMID 18959116
- [Background] Iishi H, Tatsuta M, Baba M, Uehara H, Nakaizumi A, Shinkai K, Akedo H, Funai H, Ishiguro S, Kitagawa I. Inhibition by ginsenoside Rg3 of bombesin-enhanced peritoneal metastasis of intestinal adenocarcinomas induced by azoxymethane in Wistar rats. Clin Exp Metastasis. 1997 Nov;15(6):603-11. doi: 10.1023/a:1018491314066. PMID 9344044
- [Background] Lee JY, Jung KH, Morgan MJ, Kang YR, Lee HS, Koo GB, Hong SS, Kwon SW, Kim YS. Sensitization of TRAIL-induced cell death by 20(S)-ginsenoside Rg3 via CHOP-mediated DR5 upregulation in human hepatocellular carcinoma cells. Mol Cancer Ther. 2013 Mar;12(3):274-85. doi: 10.1158/1535-7163.MCT-12-0054. Epub 2012 Oct 10. PMID 23053497
- [Background] Zhang C, Liu L, Yu Y, Chen B, Tang C, Li X. Antitumor effects of ginsenoside Rg3 on human hepatocellular carcinoma cells. Mol Med Rep. 2012 May;5(5):1295-8. doi: 10.3892/mmr.2012.808. Epub 2012 Feb 23. PMID 22366885
- [Background] Park HM, Kim SJ, Kim JS, Kang HS. Reactive oxygen species mediated ginsenoside Rg3- and Rh2-induced apoptosis in hepatoma cells through mitochondrial signaling pathways. Food Chem Toxicol. 2012 Aug;50(8):2736-41. doi: 10.1016/j.fct.2012.05.027. Epub 2012 May 22. PMID 22634290